CLINICAL TRIAL: NCT03139552
Title: Influence of Food Liking of Adding Spices to Replace Dietary Sugar Using Sequential Monadic CLT Methodology
Brief Title: Influence on Food Liking of Adding Spices to Replace Sugar Using CLT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: McCormick Science Institute (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 16-1599
Record Dates: First submitted 2017-04-26; First posted 2017-05-04 (Actual); Results first posted 2018-11-02 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2018-03

CONDITIONS: Normal Subjects Who Agree to Participate in Taste Testing
Keywords: Taste Test; Spices; Reduced sugar; Food liking
MeSH Terms: interventions — Tea

STUDY DESIGN:
Intervention Model Description: Subjects were asked to taste test 3 versions of test items (in randomized order) and provide a liking score for each.
Who Masked: Participant
Masking Description: Subjects were blind to the differences in recipes when taste testing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- full sugar recipe (Active Comparator): Each subject was randomly assigned to one of six possible sequences to taste three recipes of each test item (apple crisp, tea and oatmeal). The three recipes were full sugar recipe (FS), reduced sugar recipe (RS) and reduced sugar plus spice recipe (RSS). Each subject was randomly assigned to one of the below sequence schedules for each taste test whereby A, B, and C refer to one of the three recipes (FS, RS, or RSS):
  Sequence 1: A, B, C Sequence 2: A, C, B Sequence 3: B, A, C Sequence 4: B, C, A Sequence 5: C, A, B Sequence 6: C, B, A
  Interventions: Other: Apple Crisp; Other: Tea; Other: Oatmeal
- reduced sugar recipe (Experimental): Each subject was randomly assigned to one of six possible sequences to taste three recipes of each test item (apple crisp, tea and oatmeal). The three recipes were full sugar recipe (FS), reduced sugar recipe (RS) and reduced sugar plus spice recipe (RSS). Each subject was randomly assigned to one of the below sequence schedules for each taste test whereby A, B, and C refer to one of the three recipes (FS, RS, or RSS):
  Sequence 1: A, B, C Sequence 2: A, C, B Sequence 3: B, A, C Sequence 4: B, C, A Sequence 5: C, A, B Sequence 6: C, B, A
  Interventions: Other: Apple Crisp; Other: Tea; Other: Oatmeal
- reduced sugar plus spice recipe (Experimental): Each subject was randomly assigned to one of six possible sequences to taste three recipes of each test item (apple crisp, tea and oatmeal). The three recipes were full sugar recipe (FS), reduced sugar recipe (RS) and reduced sugar plus spice recipe (RSS). Each subject was randomly assigned to one of the below sequence schedules for each taste test whereby A, B, and C refer to one of the three recipes (FS, RS, or RSS):
  Sequence 1: A, B, C Sequence 2: A, C, B Sequence 3: B, A, C Sequence 4: B, C, A Sequence 5: C, A, B Sequence 6: C, B, A
  Interventions: Other: Apple Crisp; Other: Tea; Other: Oatmeal

INTERVENTIONS:
Other: Apple Crisp — Subjects tasted the three recipes (full sugar recipe, reduced sugar recipe, and reduced sugar plus spice recipe) of apple crisp in a randomized sequence schedule. Tastings for each test item (apple crisp, tea and oatmeal) were done during separate weeks. Subjects tasted each recipe of an item at one sitting (ie: subject completed apple crisp tastings during one seating during first week, oatmeal tastings during one seating the next week and tea tastings during one seating the next and final week).
Other: Tea — Subjects tasted the three recipes (full sugar recipe, reduced sugar recipe, and reduced sugar plus spice recipe) of tea in a randomized sequence schedule. Tastings for each test item (apple crisp, tea and oatmeal) were done during separate weeks. Subjects tasted each recipe of an item at one sitting (ie: subject completed apple crisp tastings during one seating during first week, oatmeal tastings during one seating the next week and tea tastings during one seating the next and final week).
Other: Oatmeal — Subjects tasted the three recipes (full sugar recipe, reduced sugar recipe, and reduced sugar plus spice recipe of oatmeal in a randomized sequence schedule. Tastings for each test item (apple crisp, tea and oatmeal) were done during separate weeks. Subjects tasted each recipe of an item at one sitting (ie: subject completed apple crisp tastings during one seating during first week, oatmeal tastings during one seating the next week and tea tastings during one seating the next and final week).

SUMMARY:
This study aims to reduce the amount of sugar in a particular food item and add spices to see if the food liking of that item rates as high or higher in a post meal survey. Through taste testing of the menu items (using sequential monadic CLT methodology) the investigators will determine an opinion of the participants. Results of these surveys will determine whether participants enjoy the reduced sugar options as much as their full sugar counterparts.

DETAILED DESCRIPTION:
The investigators will compare the overall consumer acceptability of each of three test items (tea, oatmeal and apple crisp) across the three test conditions using central location test (CLT) and cross-over design. The three test conditions for each test item will be (1) Full sugar ("FS"), (2) reduced sugar (and calorie) with no added spice ("RS") and (3) reduced sugar (and calorie) plus spice ("RSS"). The two reduced sugar items will be matched for calories. Subjects will be provided the test items using sequential monadic CLT methodology (Central Location Test methodology which involves product evaluation after a brief exposure (one sample-subject contact) under standardized conditions whereby subjects are given each of the 3 recipes of each test item (e.g., oatmeal with full sugar, oatmeal with reduced sugar, oatmeal with reduced plus spice) back to back (all within one sitting) in a random order. The investigators are interested in using the sequential monadic CLT methodology and having subjects taste all 3 recipes of each item in one sitting which is a commonly used test modality for sensory studies.

ELIGIBILITY:
Inclusion Criteria:

-ages 18-65

Exclusion Criteria:

* diagnosed taste or sensory disorder
* known eating disorder
* allergies to test food/ingredients
* medical conditions that may adversely affect taste (ie: dysgeusia)
* inability to complete protocol or to participate in all three taste testing sessions
* personal dietary restrictions towards test items
* dislike of the particular food items to be served in taste tests
* subjects who do not consume foods or beverages that contain sugar or to which they have added sugar will be excluded
* subjects who have not consumed or would not be willing to consume hot tea, oatmeal or baked apple products will be excluded
* subjects who are pregnant or trying to become pregnant will be excluded

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-10-17 (Actual); Primary Completion 2016-12-09 (Actual); Study Completion 2016-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John C. Peters, PhD, Principal Investigator — University of Colorado, Denver

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Krauss RM, Eckel RH, Howard B, Appel LJ, Daniels SR, Deckelbaum RJ, Erdman JW Jr, Kris-Etherton P, Goldberg IJ, Kotchen TA, Lichtenstein AH, Mitch WE, Mullis R, Robinson K, Wylie-Rosett J, St Jeor S, Suttie J, Tribble DL, Bazzarre TL. AHA Dietary Guidelines: revision 2000: A statement for healthcare professionals from the Nutrition Committee of the American Heart Association. Circulation. 2000 Oct 31;102(18):2284-99. doi: 10.1161/01.cir.102.18.2284. No abstract available. PMID 11056107
- [Background] Essed NH, Kleikers S, van Staveren WA, Kok FJ, de Graaf C. No effect on intake and liking of soup enhanced with mono-sodium glutamate and celery powder among elderly people with olfactory and/or gustatory loss. Int J Food Sci Nutr. 2009;60 Suppl 5:143-54. doi: 10.1080/09637480802710216. Epub 2009 May 21. PMID 19462326
- [Background] Howard BV, Wylie-Rosett J. Sugar and cardiovascular disease: A statement for healthcare professionals from the Committee on Nutrition of the Council on Nutrition, Physical Activity, and Metabolism of the American Heart Association. Circulation. 2002 Jul 23;106(4):523-7. doi: 10.1161/01.cir.0000019552.77778.04. No abstract available. PMID 12135957
- [Background] Trumbo P, Schlicker S, Yates AA, Poos M; Food and Nutrition Board of the Institute of Medicine, The National Academies. Dietary reference intakes for energy, carbohydrate, fiber, fat, fatty acids, cholesterol, protein and amino acids. J Am Diet Assoc. 2002 Nov;102(11):1621-30. doi: 10.1016/s0002-8223(02)90346-9. No abstract available. PMID 12449285
- [Background] Johnson RJ, Segal MS, Sautin Y, Nakagawa T, Feig DI, Kang DH, Gersch MS, Benner S, Sanchez-Lozada LG. Potential role of sugar (fructose) in the epidemic of hypertension, obesity and the metabolic syndrome, diabetes, kidney disease, and cardiovascular disease. Am J Clin Nutr. 2007 Oct;86(4):899-906. doi: 10.1093/ajcn/86.4.899. PMID 17921363
- [Background] King, SC, Snow, J, Meiselman, HL, Sainsbury, J, Carr, BT, McCafferty, D, Serrano, D, Gillette, M, Millard, L, Li, Q. Development of a questionnaire to measure consumer wellness associated with foods; The WellSense Profile. Food Quality and Preference 39: 82-94, 2014.
- [Background] Littell, RC, Miliken, GA, Stroup, WW, Wolfinger, RD, Schabenberger, O (eds.). SAS for Mixed Models, Second edn. Car, NC: SAS Institute Inc.; 2006.
- [Background] Malik VS, Popkin BM, Bray GA, Despres JP, Hu FB. Sugar-sweetened beverages, obesity, type 2 diabetes mellitus, and cardiovascular disease risk. Circulation. 2010 Mar 23;121(11):1356-64. doi: 10.1161/CIRCULATIONAHA.109.876185. No abstract available. PMID 20308626
- [Background] Peters JC, Polsky S, Stark R, Zhaoxing P, Hill JO. The influence of herbs and spices on overall liking of reduced fat food. Appetite. 2014 Aug;79:183-8. doi: 10.1016/j.appet.2014.04.019. Epub 2014 Apr 24. PMID 24769295
- [Background] Polsky S, Beck J, Stark RA, Pan Z, Hill JO, Peters JC. The influence of herbs, spices, and regular sausage and chicken consumption on liking of reduced fat breakfast and lunch items. J Food Sci. 2014 Oct;79(10):S2117-26. doi: 10.1111/1750-3841.12643. Epub 2014 Sep 12. PMID 25219391
- [Background] McGuire S. U.S. Department of Agriculture and U.S. Department of Health and Human Services, Dietary Guidelines for Americans, 2010. 7th Edition, Washington, DC: U.S. Government Printing Office, January 2011. Adv Nutr. 2011 May;2(3):293-4. doi: 10.3945/an.111.000430. Epub 2011 Apr 30. No abstract available. PMID 22332062
- [Result] Peters JC, Marker R, Pan Z, Breen JA, Hill JO. The Influence of Adding Spices to Reduced Sugar Foods on Overall Liking. J Food Sci. 2018 Mar;83(3):814-821. doi: 10.1111/1750-3841.14069. Epub 2018 Feb 24. PMID 29476623

RESULTS

PARTICIPANT FLOW:
Groups:
- Taste Testers: 150 subjects were enrolled to participate in three taste test sessions of apple crisp, tea and oatmeal. At each session, three recipes of each item were tasted. Each subject was randomly assigned to one of six possible sequences to taste the three recipes. The three recipes were full sugar recipe (FS), reduced sugar recipe (RS) and reduced sugar plus spice recipe (RSS). Each subject was randomly assigned to one of the below sequence schedules for each taste test whereby A, B, and C refer to one of the three recipes (FS, RS, or RSS): Sequence 1: A, B, C Sequence 2: A, C, B Sequence 3: B, A, C Sequence 4: B, C, A Sequence 5: C, A, B Sequence 6: C, B, A
  Subjects tasted the three recipes (full sugar recipe, reduced sugar recipe, and reduced sugar plus spice recipe) of each item in a randomized sequence schedule. Tastings for each test item (apple crisp, tea and oatmeal) were done during separate weeks. Subjects tasted all three recipes of an item at one sitting.
Period: Overall Study
Arm/Group | Taste Testers
Started | 150
Completed (3 subjects did not complete tastings of all three items.) | 147
Not Completed | 3
Not completed — unable to attend tasting due to schedule | 3

BASELINE CHARACTERISTICS:
Groups:
- Taste Testers: 150 subjects were enrolled to taste three recipes of apple crisp, tea and oatmeal. Subjects were asked to paricitpate in tastings of all three items.Each subject was randomly assigned to one of six possible sequences to taste three recipes of each test item (apple crisp, tea and oatmeal). The three recipes were full sugar recipe (FS), reduced sugar recipe (RS) and reduced sugar plus spice recipe (RSS). Each subject was randomly assigned to one of the below sequence schedules for each taste test whereby A, B, and C refer to one of the three recipes (FS, RS, or RSS): Sequence 1: A, B, C Sequence 2: A, C, B Sequence 3: B, A, C Sequence 4: B, C, A Sequence 5: C, A, B Sequence 6: C, B, A
  Taste testings ofeach test item (apple crisp, tea and oatmeal) were done during separate weeks. Subjects tasted all three recipes of an item at one sitting (ie: subject completed apple crisp tastings during one seating during first week).
Arm/Group | Taste Testers
Number analyzed (Participants) | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.9 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 118
  Male | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16
  Not Hispanic or Latino | 114
  Unknown or Not Reported | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 18
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 7
  White | 119
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 150

OUTCOME MEASURES:

1. Primary Outcome: Overall Liking of Apple Crisp
Description: Overall liking of apple crisp with a 9-point hedonic rating scale instrument (whereby 0 = dislike extremely and 9 = like extremely )
Time Frame: Day of taste testing
Measure: Mean (Standard Deviation); unit: score on likert rating scale
Groups:
- Full Sugar Recipe; Reduced Sugar Recipe; Reduced Sugar Plus Spice Recipe: Each subject was randomly assigned to one of six possible sequences to taste three recipes of each test item (apple crisp, tea and oatmeal). The three recipes were full sugar recipe (FS), reduced sugar recipe (RS) and reduced sugar plus spice recipe (RSS). Each subject was randomly assigned to one of the below sequence schedules for each taste test whereby A, B, and C refer to one of the three recipes (FS, RS, or RSS):
  Sequence 1: A, B, C Sequence 2: A, C, B Sequence 3: B, A, C Sequence 4: B, C, A Sequence 5: C, A, B Sequence 6: C, B, A
  Subjects tasted the three recipes (full sugar recipe, reduced sugar recipe, and reduced sugar plus spice recipe) of each item in a randomized sequence schedule. Tastings for each test item (apple crisp, tea and oatmeal) were done during separate weeks. Subjects tasted each recipe of an item at one sitting.
Arm/Group | Full Sugar Recipe | Reduced Sugar Recipe | Reduced Sugar Plus Spice Recipe
Number analyzed (Participants) | 150 | 150 | 150
score on likert rating scale | 7.31 (1.23) | 6.83 (1.25) | 7.22 (1.37)

2. Primary Outcome: Overall Liking of Tea
Description: Overall liking of tea with a 9-point hedonic rating scale instrument (whereby 0 = dislike extremely and 9 = like extremely )
Time Frame: day of taste testing
Measure: Mean (Standard Deviation); unit: score on a likert rating scale
Arm/Group | Full Sugar Recipe | Reduced Sugar Recipe | Reduced Sugar Plus Spice Recipe
Number analyzed (Participants) | 149 | 149 | 149
score on a likert rating scale | 6.00 (1.64) | 5.62 (1.81) | 5.85 (1.82)

3. Primary Outcome: Overall Liking of Oatmeal
Description: Overall liking of oatmeal with a 9-point hedonic rating scale instrument (whereby 0 = dislike extremely and 9 = like extremely )
Time Frame: day of taste testing
Measure: Mean (Standard Deviation); unit: score on a likert rating scale
Arm/Group | Full Sugar Recipe | Reduced Sugar Recipe | Reduced Sugar Plus Spice Recipe
Number analyzed (Participants) | 148 | 148 | 148
score on a likert rating scale | 6.84 (1.49) | 5.70 (1.45) | 6.15 (1.54)

4. Secondary Outcome: Ranking of Full Sugar Recipe of Apple Crisp
Description: Subjects ranked each recipe in order of likability as first, second or third.
Time Frame: day of taste testing
Measure: Count of Participants; unit: Participants
Groups:
- First Place Ranking: Number of subjects who rated this recipe in first place (most likable)
- Second Place Ranking: Number of subjects who rated this recipe in second place
- Third Place Ranking: Number of subjects who rated this recipe in third place (least likable)
Arm/Group | First Place Ranking | Second Place Ranking | Third Place Ranking
Number analyzed (Participants) | 150 | 150 | 150
Participants | 54 | 63 | 33

5. Secondary Outcome: Ranking of Reduced Sugar Recipe of Apple Crisp
Description: Subjects ranked each recipe in order of likability as first, second or third.
Time Frame: day of taste testing
Measure: Count of Participants; unit: Participants
Arm/Group | First Place Ranking | Second Place Ranking | Third Place Ranking
Number analyzed (Participants) | 150 | 150 | 150
Participants | 33 | 43 | 74

6. Secondary Outcome: Ranking of Reduced Sugar Plus Spice Recipe of Apple Crisp
Description: Subjects ranked each recipe in order of likability as first, second or third.
Time Frame: day of taste testing
Measure: Count of Participants; unit: Participants
Arm/Group | First Place Ranking | Second Place Ranking | Third Place Ranking
Number analyzed (Participants) | 150 | 150 | 150
Participants | 63 | 44 | 43

7. Secondary Outcome: Ranking of Reduced Sugar Recipe of Tea
Description: Subjects ranked each recipe in order of likability as first, second or third.
Time Frame: Day of taste testings
Measure: Count of Participants; unit: Participants
Arm/Group | First Place Ranking | Second Place Ranking | Third Place Ranking
Number analyzed (Participants) | 149 | 149 | 149
Participants | 34 | 58 | 57

8. Secondary Outcome: Ranking of Full Sugar Recipe of Tea
Description: Subjects ranked each recipe in order of likability as first, second or third.
Time Frame: day of taste testing
Measure: Count of Participants; unit: Participants
Arm/Group | First Place Ranking | Second Place Ranking | Third Place Ranking
Number analyzed (Participants) | 149 | 149 | 149
Participants | 66 | 41 | 42

9. Secondary Outcome: Ranking of Reduced Sugar Plus Spice Recipe of Tea
Description: Subjects ranked each recipe in order of likability as first, second or third.
Time Frame: day of taste testing
Measure: Count of Participants; unit: Participants
Arm/Group | First Place Ranking | Second Place Ranking | Third Place Ranking
Number analyzed (Participants) | 149 | 149 | 149
Participants | 49 | 50 | 50

10. Secondary Outcome: Ranking of Reduced Sugar Recipe of Oatmeal
Description: Subjects ranked each recipe in order of likability as first, second or third.
Time Frame: day of taste testing
Measure: Count of Participants; unit: Participants
Arm/Group | First Place Ranking | Second Place Ranking | Third Place Ranking
Number analyzed (Participants) | 148 | 148 | 148
Participants | 12 | 49 | 87

11. Secondary Outcome: Ranking of Full Sugar Recipe of Oatmeal
Description: Subjects ranked each recipe in order of likability as first, second or third.
Time Frame: day of taste testing
Measure: Count of Participants; unit: Participants
Arm/Group | First Place Ranking | Second Place Ranking | Third Place Ranking
Number analyzed (Participants) | 148 | 148 | 148
Participants | 88 | 39 | 21

12. Secondary Outcome: Ranking of Reduced Sugar Plus Spice Oatmeal
Description: Subjects ranked each recipe in order of likability as first, second or third.
Time Frame: day of taste testing
Measure: Count of Participants; unit: Participants
Arm/Group | First Place Ranking | Second Place Ranking | Third Place Ranking
Number analyzed (Participants) | 148 | 148 | 148
Participants | 48 | 60 | 40

ADVERSE EVENTS:
Description: Information on adverse events was not collected; subjects were not queried about whether they experienced any adverse events. No subjects reported any adverse events during the study.
Groups:
- Full Sugar Recipe; Reduced Sugar Recipe; Reduced Sugar Plus Spice Recipe: Each subject was randomly assigned to one of six possible sequences to taste three recipes of each test item (apple crisp, tea and oatmeal). The three recipes were full sugar recipe (FS), reduced sugar recipe (RS) and reduced sugar plus spice recipe (RSS). Each subject was randomly assigned to one of the below sequence schedules for each taste test whereby A, B, and C refer to one of the three recipes (FS, RS, or RSS):
  Sequence 1: A, B, C Sequence 2: A, C, B Sequence 3: B, A, C Sequence 4: B, C, A Sequence 5: C, A, B Sequence 6: C, B, A
  Apple Crisp: Subjects tasted the three recipes (full sugar recipe, reduced sugar recipe, and reduced sugar plus spice recipe) of apple crisp in a randomized sequence schedule. Tastings for each test item (apple crisp, tea and oatmeal) were done during separate weeks. Subjects tasted each recipe of an item at one sitting.
Arm/Group | Full Sugar Recipe | Reduced Sugar Recipe | Reduced Sugar Plus Spice Recipe
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Due to the nature of the study involving different food recipes, the food preparation staff were not blinded to treatment. The participants were blinded to treatment. Therefore, the study was single blind.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No